CLINICAL TRIAL: NCT03235570
Title: A Phase 1, Open-Label, Dose-Escalation, Dose-Expansion, Safety and Tolerability Study of Pemigatinib in Japanese Subjects With Advanced Malignancies - (FIGHT-102)
Brief Title: A Safety and Tolerability Study of Pemigatinib in Japanese Subjects With Advanced Malignancies - (FIGHT-102)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 54828-102
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Solid Tumors
Keywords: Solid tumor; malignancy; fibroblast growth factor receptor (FGFR); fibroblast growth factor (FGF)/FGFR alteration
MeSH Terms: conditions — Neoplasms; Acrocephalosyndactylia | interventions — pemigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pemigatinib (Experimental): Part 1 is an open-label dose-escalation design based on observing each dose level for a period of 21 days. Part 2 will evaluate the recommended dose determined in Part 1.
  Interventions: Drug: Pemigatinib

INTERVENTIONS:
Drug: Pemigatinib — Pemigatinib at the protocol-defined dose administered once daily.
  Other Names: INCB054828

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of pemigatinib in Japanese subjects with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

* First generation Japanese; subject was born in Japan and has not lived outside of Japan for a total of > 10 years and subject can trace maternal and paternal Japanese ancestry.
* Part 1: Any histologically confirmed advanced solid tumor malignancy. Subjects enrolled at a lower dose level expansion cohort are required to have documented FGF/FGFR alterations and baseline and on-treatment tumor biopsy for testing of biomarkers.
* Part 2: Any histologically confirmed advanced solid tumor malignancy with a FGF/FGFR alteration
* Advanced or metastatic and recurrent cancer where an appropriate treatment option is not available.
* Life expectancy > 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status: Part 1: 0 or 1; Part 2: 0, 1, or 2.
* Genomic testing is mandatory for all enrolled subjects. Archival tumor specimen of at least 7 slides or willingness to undergo a pretreatment tumor biopsy to provide a tumor block or at least 7 unstained slides. Archival tumor biopsies are acceptable at baseline and should be no more than 2 years old (preferably less than 1 year old and collected since the completion of the last treatment); subjects with samples older than 2 years old and/or with sequencing report from the central laboratory require approval from the sponsor medical monitor for exemption from tumor biopsy or tumor sample requirement.

Exclusion Criteria:

* Treatment with other investigational study drug for any indication for any reason, or receipt of anticancer medications within 21 days or 5 half-lives (whichever is longer) before first dose of study drug (6 weeks for mitomycin-C or nitrosoureas, 7 days for tyrosine kinase inhibitors).
* Prior receipt of a selective FGFR inhibitor.
* Laboratory and medical history parameters outside Protocol-defined range.
* History and/or current evidence of ectopic mineralization/calcification including but not limited to soft tissue, kidneys, intestine, myocardia, or lung, excepting calcified lymph nodes and asymptomatic arterial or cartilage/tendon calcification.
* Current evidence of corneal disorder/keratopathy including but not limited to bullous/band keratopathy, corneal abrasion, inflammation/ulceration, keratoconjunctivitis, confirmed by ophthalmologic examination.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed by monitoring frequency, duration, and severity of adverse events (AEs) | Baseline through 30 days after end of treatment, up to approximately 16 months.
  An AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurs after a subject provides informed consent.

SECONDARY OUTCOMES:
Overall response rate in subjects with measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Baseline and Day 15 of every third treatment cycle, up to approximately 6 months
  Defined as proportion of subjects who meet the response criteria (complete response + partial response) as appropriate for the tumor type.
Pharmacodynamics of pemigatinib assessed by changes in serum phosphorus level | Baseline and protocol-defined timepoints throughout the treatment period, up to approximately 6 months
  Analyzed to look for differences that may be associated with response or safety as well as significant changes associated with treatment.
Observed Plasma Concentration of pemigatinib | During the first cycle, up to Day 16
  PK parameters will be calculated from the blood plasma concentrations of pemigatinib using standard noncompartmental (model independent) PK methods.

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterine Asatiani, MD, Study Director — Incyte Corporation
Locations (12):
- Japan (12):
  - Aichi Cancer Center Hospital, Aichi
  - Chiba Cancer Center, Chiba
  - National Cancer Central Hospital East, Chiba
  - Kyusyu Cancer Center, Fukuoka
  - Kanazawa University Hospital, Ishikawa
  - Kanagawa Cancer Center, Kanagawa
  - Osaka International Cancer Institute, Osaka
  - Saitama Cancer Center, Saitama
  - Hokkaido Cancer Center, Sapporo
  - Shizuoka Cancer Center, Shizuoka
  - National Cancer Central Hospital, Tokyo
  - JFCR Ariake Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No